CLINICAL TRIAL: NCT04314713
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Dose-Escalation Study To Evaluate The Safety, Tolerability, and Pharmacokinetics Of Intramuscular Administration Of Scopolamine Hydrobromide Trihydrate, Injection
Brief Title: A Study to Evaluate the Intramuscular Administration of Scopolamine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: DSMB decision due to adverse events
Sponsor: Battelle Memorial Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S-16-14
Record Dates: First submitted 2020-03-10; First posted 2020-03-19 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Medical Countermeasures; Organophosphate Poisoning
Keywords: Scopolamine
MeSH Terms: conditions — Organophosphate Poisoning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded, randomized, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Scopolamine HBT 0.005 mg/kg (Placebo Comparator): Dose of Scopolamine 0.005mg/kg verses Placebo
  Interventions: Drug: Scopolamine Hydrobromide Trihydrate
- Scopolamine HBT 0.007 mg/kg (Placebo Comparator): Dose of Scopolamine 0.007mg/kg verses Placebo
  Interventions: Drug: Scopolamine Hydrobromide Trihydrate
- Scopolamine HBT 0.011 mg/kg (Placebo Comparator): Dose of Scopolamine 0.011mg/kg verses Placebo
  Interventions: Drug: Scopolamine Hydrobromide Trihydrate
- Scopolamine HBT 0.014 mg/kg (Placebo Comparator): Dose of Scopolamine 0.014mg/kg verses Placebo
  Interventions: Drug: Scopolamine Hydrobromide Trihydrate
- Scopolamine HBT 0.021 mg/kg (Placebo Comparator): Dose of Scopolamine 0.021mg/kg verses Placebo
  Interventions: Drug: Scopolamine Hydrobromide Trihydrate
- Placebo (No Intervention): Placebo controlled

INTERVENTIONS:
Drug: Scopolamine Hydrobromide Trihydrate — Scopolamine Hydrobromide Trihydrate Intramuscular Injection
  Arms: Scopolamine HBT 0.005 mg/kg; Scopolamine HBT 0.007 mg/kg; Scopolamine HBT 0.011 mg/kg; Scopolamine HBT 0.014 mg/kg; Scopolamine HBT 0.021 mg/kg

SUMMARY:
To characterize the safety and tolerability profile of ascending doses of scopolamine hydrobromide trihydrate (Scopolamine HBT) administered by intramuscular (IM) injection. And characterize the pharmacokinetics (PK) of ascending doses of Scopolamine HBT administered by IM injection

DETAILED DESCRIPTION:
This is a double-blinded, randomized, placebo-controlled, in-clinic, Phase 1, single-dose, IM, sequential dose-escalation study in healthy adults aged 18-55. Healthy volunteers will be assigned to 1 of 5 cohorts of Scopolamine HBT dosage groups: 0.005, 0.007, 0.011, 0.014, or 0.021 mg/kg, or will receive the placebo administered by IM injection to the anterior thigh. In each cohort, 6 to 9 subjects will receive active drug and 2 to 3 subjects will receive placebo. Each cohort will have at least 3 male and 3 female subjects enrolled among the first 8 subjects in the dosing group to ensure that at least 1 male subject and 1 female subject in each dosing group receive active drug. If nonextreme dose-limiting toxicities are observed in any of the cohorts, 4 additional subjects, 3 active and 1 placebo, may be added to each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 55 years of age, inclusive, at the time of drug administration
2. Without clinically significant abnormities on physical examination at screening or prior to drug administration
3. Generally healthy, as determined by medical history review, physical examination, and laboratory testing at screening and prior to drug administration
4. Must have a BMI (body mass index) of ≥ 19.0 and ≤ 30.0, and weight range of 55.0 to 85.0 kg at screening or prior to drug administration
5. Must have adequate venous access and sufficient upper leg muscle tissue for drug administration
6. If female, the subject must be nonpregnant and nonbreastfeeding, and have a negative serum pregnancy test at screening and prior to drug administration
7. If female of childbearing potential, the subject must have been using adequate contraception (as defined in Section 5.3.1.5) for at least 3 months prior to drug administration and must agree to use an adequate method of contraception for at least 30 days following drug administration
8. Females of nonchildbearing potential are also eligible, defined as a subject who is postmenopausal (continuous amenorrhea for 24 months) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy)
9. A male with a female partner of childbearing potential must agree to use a barrier method of contraception (defined as condoms with spermicide) for at least 30 days following drug administration
10. If male, must not have past diagnoses of benign prostatic hypertrophy or urinary tract obstruction and must not have on screening history/review of systems symptoms suggestive of urinary tract obstruction (eg, urinary hesitancy, urgency, frequency, or nocturia)
11. Nonsmoker/tobacco/nicotine product (including e-cigarettes) user within 3 months of first dosing and must have a total lifetime exposure to cigarettes of < 15 pack-years
12. No evidence of significant neuropsychiatric disorders based on the Brief Psychiatric Rating Scale (BPRS) at screening and prior to drug administration, which is defined as having a global score of ≤ 25 with no score higher than 2 on any one item, with the exception of a score of 1 (ie, Not Present) to disorientation, hallucinatory behavior, and suspiciousness (ie, paranoia)
13. No evidence of suicidal ideation or behavior at screening and prior to drug administration, which is defined as having a global score of 0 on the Columbia-Suicide Severity Rating Scale (C-SSRS)
14. Ability to read, speak, and comprehend English and a willingness to sign informed consent

Exclusion Criteria:

1. Received any other investigational drug within 30 days prior to drug administration
2. Known allergies to any component of the study drug, other belladonna alkaloids, or the recovery medications (physostigmine, atropine, or benzodiazepines [diazepam or lorazepam])
3. History of migraine headaches or seizures
4. History of psychosis or psychotic episodes
5. Clinically relevant abnormal physical findings (including vital signs) as determined by the investigator at screening or prior to drug administration that could interfere with the objectives of the study or the safety of the subject
6. Has ongoing drug abuse/dependence (including alcohol), recent history (over the past 5 years) of treatment for alcohol or drug abuse, or a current positive alcohol breathalyzer test or current positive urine test for drugs of abuse (as defined in Section 11.1.9.5) at screening or prior to drug administration
7. Has consumed Seville orange (bitter orange), grapefruit, grapefruit juice, other grapefruit-containing products, or starfruit within 7 days prior to dosing
8. Has consumed caffeine or other xanthine-containing products within 7 days prior to dosing
9. Has any specified laboratory values (eg, hematology, serum chemistry, and urinalysis) outside of the normal range for age and sex and deemed clinically significant by the investigator within 30 days before drug administration
10. Has positive (reactive) test results for hepatitis B surface antigen, hepatitis C, syphilis, HIV-1, or HIV-2
11. Has narrow-angle glaucoma or high intraocular pressures in either or both eyes
12. Has pyloric obstruction or urinary bladder neck obstruction
13. Has impaired liver or kidney functions
14. Clinically relevant electrocardiogram (ECG) abnormalities on any 12-lead ECG obtained at screening or prior to dosing
15. ECG with a PR interval ≥ 200 msec at screening or prior to dosing
16. ECG with QRS duration > 120 msec at screening or prior to dosing
17. ECG RR interval > 1500 msec at screening or prior to dosing
18. ECG with a QTc interval > 450 msec for males or 470 msec for females (QT interval corrected with Fridericia correction [QTcF]) at screening or prior to dosing
19. Systolic blood pressure > 140 mm Hg and/or diastolic blood pressure > 90 mm Hg at screening or prior to dosing
20. Systolic blood pressure < 90 mm Hg and/or diastolic blood pressure < 50 mm Hg at screening or prior to dosing
21. Currently taking or has taken other antimuscarinic drugs such as phenothiazines, tricyclic antidepressants, antihistamines (including meclizine), meperidine, or other anticholinergics that have weak antimuscarinic activity or that cause drowsiness, including antidepressants, benzodiazepines, alcohol, sedatives (used to treat insomnia), pain relievers, anxiety medicines, and muscle relaxants within 72 hours prior to dosing
22. Has taken, within 14 days of planned dosing, any prescription or nonprescription medication (including home remedies, herbal supplements, or nutritional supplements) unless the PI/subinvestigator, in consultation with the medical monitor, provides a statement justifying that the medication taken will not impact the results of this study (with rare exceptions taking prescriptions drugs will be grounds for exclusion)
23. History of major DSM-5 Axis I or II disorder, or evidence of such disorder at Day -1 as determined via the Structured Clinical Interview for DSM-5, customized Clinical Trials version (SCID-5-CT)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo DePetrillo, MD, Principal Investigator — Pharmaron
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Scopolamine HBT 0.005 mg/kg: IM Dose of Scopolamine 0.005mg/kg verses Placebo once on Day 1
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 2 Scopolamine HBT 0.007 mg/kg: IM Dose of Scopolamine 0.007mg/kg verses Placebo once on Day 1
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 3 Scopolamine HBT 0.011 mg/kg: IM Dose of Scopolamine 0.011mg/kg verses Placebo once on Day 1
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 4 Scopolamine HBT 0.014 mg/kg: IM Dose of Scopolamine 0.014mg/kg verses Placebo once on Day 1
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 5 Scopolamine HBT 0.021 mg/kg: IM Dose of Scopolamine 0.021mg/kg verses Placebo once on Day 1
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
Period: Overall Study
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg | Cohort 5 Scopolamine HBT 0.021 mg/kg | Placebo
Started | 6 | 6 | 6 | 6 | 0 (On 13 June 2021, following DSMB recommendation and final sponsor decision, the PI was notified of the sponsor's decision to close the study to enrollment and not proceed to Cohort 5 (0.021 mg/kg).) | 8
Completed | 6 | 6 | 6 | 5 | 0 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: On 13 June 2021, following DSMB recommendation and final sponsor decision, the PI was notified of the sponsor's decision to close the study to enrollment and not proceed to Cohort 5 (0.021 mg/kg).
Groups:
- Cohort 1 Scopolamine HBT 0.005 mg/kg: Dose of Scopolamine 0.005mg/kg verses Placebo
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 2 Scopolamine HBT 0.007 mg/kg: Dose of Scopolamine 0.007mg/kg verses Placebo
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 3 Scopolamine HBT 0.011 mg/kg: Dose of Scopolamine 0.011mg/kg verses Placebo
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 4 Scopolamine HBT 0.014 mg/kg: Dose of Scopolamine 0.014mg/kg verses Placebo
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Cohort 5 Scopolamine HBT 0.021 mg/kg: Dose of Scopolamine 0.021mg/kg verses Placebo
  Scopolamine Hydrobromide Trihydrate: Scopolamine Hydrobromide Trihydrate Intramuscular Injection
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg | Cohort 5 Scopolamine HBT 0.021 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 8 | 32
Age, Customized [Mean (Standard Deviation); unit: years] — 18 to 55 years of age
  years
    Age (years) mean | 34.8 (9.6) | 34.8 (9.11) | 31.7 (10.31) | 35.7 (11.48) |  | 32.6 (10.07) | 33.8 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 2 |  | 3 | 15
  Male | 3 | 3 | 2 | 4 |  | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 2 |  | 2 | 8
  Not Hispanic or Latino | 6 | 3 | 5 | 4 |  | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 |  | 1 | 2
  Asian | 0 | 0 | 0 | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  | 0 | 0
  Black or African American | 5 | 2 | 4 | 3 |  | 5 | 19
  White | 0 | 4 | 2 | 1 |  | 2 | 9
  More than one race | 1 | 0 | 0 | 1 |  | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 |  | 8 | 32
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.55 (3.454) | 25.58 (2.143) | 24.17 (1.876) | 25.95 (2.669) |  | 24.58 (2.232) | 24.94 (2.442)

OUTCOME MEASURES:

1. Primary Outcome: Determine Degree and Number of Adverse Events Experienced by Subjects.
Description: Safety and tolerability profile of ascending doses of scopolamine hydrobromide trihydrate (Scopolamine HBT) administered by intramuscular (IM) injection
Time Frame: 30 Days (+7)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg | Cohort 5 Scopolamine HBT 0.021 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 8
Participants
  Adverse Events : Subjects with at least 1 AE | 6 | 5 | 6 | 6 |  | 5
  Somnolence | 2 | 3 | 6 | 5 |  | 1
  Dizziness | 2 | 4 | 3 | 6 |  | 0
  Headache | 3 | 0 | 1 | 2 |  | 0
  Injection site pain | 1 | 2 | 2 | 2 |  | 3
  Injection site paraesthesia | 2 | 1 | 0 | 2 |  | 2
  Injection site hypoaesthesia | 1 | 0 | 1 | 2 |  | 2
  Dry mouth | 4 | 3 | 2 | 1 |  | 0
  Delirium | 0 | 0 | 0 | 3 |  | 0
  Any TEAEs | 6 | 5 | 6 | 6 |  | 5
  Any Serious TEAEs | 0 | 0 | 0 | 0 |  | 0
  Any Treatment-Related Serious TEAEs | 0 | 0 | 0 | 0 |  | 0
  Any TEAEs Leading to Discontinuation of Study Drug | 0 | 0 | 0 | 0 |  | 0
  Any TEAEs Leading to Discontinuation of Study | 0 | 0 | 0 | 0 |  | 0
  Any TEAEs Leading to Death | 0 | 0 | 0 | 0 |  | 0
  SAEs | 0 | 0 | 0 | 0 |  | 0
  DLTs | 0 | 0 | 0 | 0 |  | 0

2. Primary Outcome: Cmax of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: Cmax of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: Cmax (ug/mL)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Cmax (ug/mL) | 0.67 (0.286) | 1.07 (0.529) | 1.53 (0.501) | 1.91 (0.455)

3. Primary Outcome: Tmax of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: Tmax of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: Tmax (hr)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Tmax (hr) | 1 (0.4) | 1 (0.8) | 1 (0.6) | 1 (0.5)

4. Primary Outcome: Apparent Volume of Distribution (mL/kg) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: Apparent Volume of Distribution (mL/kg) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: Apparent Volume of Distribution (mL/kg)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Apparent Volume of Distribution (mL/kg) | 6258 (1678.1) | 5552 (1710.3) | 5963 (970.8) | 10210 (4402.5)

5. Primary Outcome: t1/2 (hr) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: t1/2 (hr) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: t1/2 (hr)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
t1/2 (hr) | 1.99 (0.235) | 1.88 (0.207) | 2.10 (0.535) | 4.47 (2.876)

6. Primary Outcome: Apparent Clearance (mL/hr/kg) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: Apparent Clearance (mL/hr/kg) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: Apparent Clearance (mL/hr/kg)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Apparent Clearance (mL/hr/kg) | 2177 (545.6) | 2100 (805.2) | 2012 (253.9) | 1765 (375.4)

7. Primary Outcome: MRT (hr) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: MRT (hr) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: MRT (hr)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
MRT (hr) | 3.18 (0.647) | 3.02 (0.639) | 3.01 (0.355) | 3.81 (0.802)

8. Primary Outcome: AUClast (hr*ug/mL) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: AUClast (hr*ug/mL) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: AUClast (hr*ug/mL)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
AUClast (hr*ug/mL) | 2.36 (0.499) | 3.67 (1.293) | 5.47 (0.694) | 8.16 (1.940)

9. Primary Outcome: AUCinfinity (hr*ug/mL) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: AUCinfinity (hr*ug/mL) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: AUCinfinity (hr*ug/mL)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
AUCinfinity (hr*ug/mL) | 2.4 (.5) | 3.7 (1.32) | 5.5 (.68) | 8.3 (1.98)

10. Primary Outcome: Cmax/Dose (ug/mL)/(mg/kg) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: Cmax/Dose (ug/mL)/(mg/kg) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: Cmax/Dose (ug/mL)/(mg/kg)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Cmax/Dose (ug/mL)/(mg/kg) | 133 (57.3) | 153 (75.6) | 139 (45.5) | 137 (32.5)

11. Primary Outcome: AUCinfinity/Dose (hr*ug/mL)/(mg/kg) of Ascending Doses of Scopolamine HBT Administered by IM Injection.
Description: AUCinfinity/Dose (hr*ug/mL)/(mg/kg) of ascending doses of Scopolamine HBT administered by IM injection.
Time Frame: 30 Days (+7)
Measure: Mean (Standard Deviation); unit: AUCinfinity/Dose (hr*ug/mL)/(mg/kg)
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
AUCinfinity/Dose (hr*ug/mL)/(mg/kg) | 481 (100.3) | 535 (188.6) | 504 (62.5) | 590 (140.4)

ADVERSE EVENTS:
Time Frame: AEs/SAEs were collected from time of dosing through 30 days (+7) after dosing.
Description: Cohort 5 number of participants affected and at risk is zero due to sponsor's decision to close the study to enrollment and not proceed to Cohort 5 (0.021 mg/kg).
Arm/Group | Cohort 1 Scopolamine HBT 0.005 mg/kg | Cohort 2 Scopolamine HBT 0.007 mg/kg | Cohort 3 Scopolamine HBT 0.011 mg/kg | Cohort 4 Scopolamine HBT 0.014 mg/kg | Cohort 5 Scopolamine HBT 0.021 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/8
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 6/6 | 6/6 | 0/0 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Scopolamine HBT 0.005 mg/kg (N=6) | Cohort 2 Scopolamine HBT 0.007 mg/kg (N=6) | Cohort 3 Scopolamine HBT 0.011 mg/kg (N=6) | Cohort 4 Scopolamine HBT 0.014 mg/kg (N=6) | Cohort 5 Scopolamine HBT 0.021 mg/kg (N=0) | Placebo (N=8)
Somnolence (Nervous system disorders) | 2 | 3 | 6 | 5 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 3 | 6 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 1 | 2 | 0 | 0
Injection site pain (General disorders) | 1 | 2 | 2 | 2 | 0 | 3
Injection site paraesthesia (General disorders) | 2 | 1 | 0 | 2 | 0 | 2
Injection site hypoaesthesia (General disorders) | 1 | 0 | 1 | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 2 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish without written authorization from the DOD.

DOCUMENTS (3):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04314713/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT04314713/SAP_001.pdf
  • Informed Consent Form (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT04314713/ICF_002.pdf